CLINICAL TRIAL: NCT06270784
Title: Traditional vs Orthodontic Extraction of Impacted Teeth Related to the Inferior Alveolar Nerve
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Marmara University (Other)
Responsible Party: Principal Investigator, Senem Askin Ekinci, Principal Investigator, Marmara University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 09.2024.122
Record Dates: First submitted 2024-02-13; First posted 2024-02-21 (Actual); Last update posted 2025-05-07 (Actual); Status verified 2024-09

CONDITIONS: Inferior Alveolar Nerve Injuries
Keywords: Mandibular nerve injuries, impacted teeth, tooth extraction
MeSH Terms: conditions — Mandibular Nerve Injuries; Tooth, Impacted

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Traditional Extraction Group (Active Comparator)
  Interventions: Procedure: Traditional Extraction
- Orthodontic Extraction Group (Experimental)
  Interventions: Procedure: Orthodontic Extraction

INTERVENTIONS:
Procedure: Traditional Extraction — Participants in this group will undergo traditional extraction method. This method involves uncovering the impacted tooth and extracting the tooth with or without dividing it.
  Arms: Traditional Extraction Group
Procedure: Orthodontic Extraction — Participants in this group will undergo orthodontic extraction method. In this method, a two-stage surgical procedure will be performed. In the first operation, the impacted tooth will be uncovered, and then a button will be placed on the tooth. For anchorage purposes, orthodontic mini screws will be placed in the mandibular ramus or zygomaticomaxillary buttress area. Elastics and/or ligature wires fixed to the button will be attached to the mini screw to provide force for the traction of the tooth.
  Patients will be called for check-up appointments every two weeks, and the movement of the impacted tooth will be monitored with panoramic x-rays. The second operation will be planned when the tooth moves away from the inferior alveolar nerve. In the second operation, the tooth will be extracted in a similar way to the traditional extraction group.
  Arms: Orthodontic Extraction Group

SUMMARY:
The aim of this clinical study was to compare the effects of traditional and orthodontic extraction methods on postoperative nerve damage in impacted third molars associated with the inferior alveolar nerve. The main question it aims to answer is:

-Does the orthodontic extraction method reduce the risk of nerve injury compared to traditional extraction?

Participants will:

* undergo either traditional or orthodontic extraction
* be monitored for postoperative paresthesia.

Researchers will compare traditional and orthodontic extraction methods to see if extraction methods affect postoperative nerve damage.

DETAILED DESCRIPTION:
The extraction of an impacted mandibular third molar is one of the most frequently performed procedures by oral and maxillofacial surgeons. The close anatomical relationship between the root of an impacted mandibular third molar and the inferior alveolar nerve may result in inferior alveolar nerve damage. The incidence of inferior alveolar nerve injury during the removal of an impacted mandibular third molar ranges from 0.35% to 8.4%. In addition to radiographic analysis, various surgical techniques, such as coronectomy, have been proposed to reduce the incidence of inferior alveolar nerve injury.

The orthodontic extraction technique is an orthodontically supported surgical approach that reduces the risk of neurological complications that may occur in inferior alveolar nerve and facilitates the surgical removal of impacted mandibular third molars close to the mandibular canal, even if they are associated with cystic lesions.

The purpose of this study is to examine the effect of orthodontic extraction applied to minimize inferior alveolar nerve damage during the extraction of deeply impacted mandibular third molar teeth on postoperative nerve injury. For this purpose, the postoperative paresthesia findings of patients who underwent orthodontic extraction will be compared with those of those who underwent traditional extraction.

ELIGIBILITY:
Inclusion Criteria:

* Presence of indication for wisdom tooth extraction for reasons such as pericoronitis, pathological formation, orthodontic reasons, caries, etc.
* Mandibular impacted wisdom teeth close to the inferior alveolar nerve

Exclusion Criteria:

* Mandibular impacted wisdom tooth not close to inferior alveolar nerve
* Wisdom tooth whose apexification has not yet been completed
* Suspicion of a malignant pathological lesion
* Pathological lesion associated with inferior alveolar nerve
* Presence of an acute infection

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 46 (Actual)
Dates: Start 2024-01-17 (Actual); Primary Completion 2024-05-06 (Actual); Study Completion 2024-11-06 (Actual)

PRIMARY OUTCOMES:
2-point discrimination test on the 7th day after surgery | A 2-point discrimination test will be performed before the extraction and 7 days after extraction in both groups.
  The primary outcome measure of the study was the assessment of nerve injury. For this purpose, postoperative nerve injury will be recorded by a 2-point discrimination test with the help of a caliper with a 1mm gap.

SECONDARY OUTCOMES:
Visual Analog Score(VAS) | VAS will be evaluated on the 7th and 14th postoperative days and the 1st, 3rd, and 6th months after tooth extraction.
  To measure the degree of nerve injury, the patient will be asked to choose a score based on the degree of numbness, where 0 indicates complete numbness and 10 indicates complete normal sensation.
2-point discrimination test on the 14th days and the 1st, 3rd, and 6th months after extraction. | A 2-point discrimation test will be performed on the 14th days and the 1st, 3rd, and 6th months after extraction.
  Nerve injury will be recorded by a 2-point discrimination test with the help of a caliper with a 1mm gap.
Inferior alveolar nerve recovery | Inferior alveolar nerve recovery will be assessed on the 7th and 14th postoperative days and the 1st, 3rd, and 6th months after tooth extraction.
  The effect of demographic data such as age, gender, and tooth position on IAN recovery will be evaluated. At postoperative time points, 2-point discrimation test values that are 2 mm more than the preoperative result will be considered to indicate nerve injury.

CONTACTS AND LOCATIONS:
Locations (1):
- Marmara University, Istanbul, Basibuyuk, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Askin Ekinci S, Kiristioglu ZB, Ates O, Gocmen G. Traditional vs. orthodontic extraction of impacted teeth related to the inferior alveolar nerve: a randomized control trial. BMC Oral Health. 2025 Jul 2;25(1):1036. doi: 10.1186/s12903-025-06402-7. PMID 40604669